CLINICAL TRIAL: NCT06970626
Title: Quality of Recovery in Laparoscopic Sleeve Gastrectomy Using Dexmedetomidine Infusion Versus Laparoscopic TAP Block in Combination With Paragastric Neural Block
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16/462
Record Dates: First submitted 2025-04-15; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Laparoscopic Sleeve Gastrectomy
Keywords: dexmedetomidine; Laparoscopic Sleeve Gastrectomy (LSG); Paragastric Neural Block; Laparoscopic TAP
MeSH Terms: interventions — Dental Occlusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group D (Active Comparator): This group (Group D) will receive intravenous loading dose of dexmedetomidine at 0.5 μg/kg ideal body weight (concentration 2 μg/ml) over 15 minutes prior to anesthesia induction, followed by 10 ml of 0.9% sodium chloride over 60 seconds during anesthetic induction. Post-intubation, Dexmedetomidine will be maintained at 0.5 μg/kg/h ideal body weight via a syringe pump until trocar removal. Paragastric neural block (PGNB) will be administered using a 25-gauge needle attached to a venous catheter extension, introduced through the left 12 mm port. Infiltration of 20 mL undiluted 0.5% bupivacaine will be performed at six levels in the fatty tissue of the paragastric area, including the lesser omentum, vagus nerve, esophago-gastric junction, proximal stomach, mid-stomach, distal antrum, hepatic artery, and left gastric artery, with the needle cap removed under direct vision throughout the procedure.
  Interventions: Drug: Dexmedetomidine infusion; Procedure: Paragastric neural block
- Group P (Active Comparator): This group (Group P) will receive Paragastric neural block (PGNB) with laparoscopic TAP block (LTAP). LTAP will be administered after insufflation before insertion of the right and left-handed ports. 30 mL of 0.25% bupivacaine will be injected into the posterolateral subcostal regions on both sides. The correct placement will be confirmed by observing the spread of fluid between the transversus abdominis and the internal oblique muscle layers laparoscopically. Paragastric neural block (PGNB) will be administered using a 25-gauge needle attached to a venous catheter extension, introduced through the left 12 mm port. Infiltration of 20 mL undiluted 0.5% bupivacaine will be performed at six levels in the fatty tissue of the paragastric area, including the lesser omentum, vagus nerve, esophago-gastric junction, proximal stomach, mid-stomach, distal antrum, hepatic artery, and left gastric artery, with the needle cap removed under direct vision throughout the procedure.
  Interventions: Procedure: Paragastric neural block; Procedure: Laparoscopic Transversus Abdominis Plane (LTAP) block

INTERVENTIONS:
Drug: Dexmedetomidine infusion — Dexmedetomidine will be maintained at 0.5 μg/kg/h ideal body weight via a syringe pump until trocar removal.
  Arms: Group D
Procedure: Paragastric neural block — Paragastric neural block (PGNB) will be administered using a 25-gauge needle attached to a venous catheter extension, introduced through the left 12 mm port. Infiltration of 20 mL undiluted 0.5% bupivacaine will be performed at six levels in the fatty tissue of the paragastric area, including the lesser omentum, vagus nerve, esophago-gastric junction, proximal stomach, mid-stomach, distal antrum, hepatic artery, and left gastric artery, with the needle cap removed under direct vision throughout the procedure.
Procedure: Laparoscopic Transversus Abdominis Plane (LTAP) block — LTAP will be administered after insufflation before insertion of the right and left-handed ports. 30 mL of 0.25% bupivacaine will be injected into the posterolateral subcostal regions on both sides. The correct placement will be confirmed by observing the spread of fluid between the transversus abdominis and the internal oblique muscle layers laparoscopically
  Arms: Group P

SUMMARY:
The goal of this clinical trial is to learn which is better, combining Dexmedetomidine infusion and paragastric neural block or combining laparoscopic TAP block and paragastric neural block to enhance recovery after laparoscopic sleeve gastrectomy.

The main questions it aims to answer are:

Will using paragastric neural block (PGNB) combined with dexmedetomidine infusion give better recovery or using PGNB combined with laparoscopic transversus abdominis plane (LTAP) block in patients undergoing laparoscopic sleeve gastrectomy.

This will be assessed by:

Recording how much opioids were consumed by the patients Hemodynamic stability of the enrolled patients Pain scores as given by the patient The quality of postoperative patient recovery How many patients encountered nausea or vomiting

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists (ASA) physical status II- III
2. BMI 35- 50 kg/m2

Exclusion Criteria:

1. Significant hepatic, renal, neuromuscular, or cardiac impairments
2. Extreme obesity (BMI > 50 kg/m2)
3. Patients on current opioid medication
4. Allergies to dexmedetomidine or bupivacaine

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2025-06-04 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Opioid Consumption | Opioid consumption will be measured at 4, 8, and 12 hours postoperatively
  Total opioids consumed by the patient will be recorded
Patient satisfaction using the QoR 40 questionnaire | Postoperative day 1
  Patient satisfaction with the procedure done will be measured using the QoR (quality of recovery)40 questionnaire. Scores range from 40 (extremely poor quality of recovery) to 200 (excellent quality of recovery)

SECONDARY OUTCOMES:
Heart Rate | Heart rate will be monitored continuously every 5 minutes and will be recorded prior to induction, post-induction, after the loading dose of dexmedetomidine, 4 hours and 12 hours postoperatively.
  Heart rate (beats/min) will be monitored continuously every 5 minutes and will be recorded prior to induction, post-induction, after the loading dose of dexmedetomidine, 4 hours and 12 hours postoperatively.
Time to mobilize | Postoperative day 1
  The time to which the patient will be able to start mobilization after surgery will be recorded (in minutes)
Incidence of nausea and vomiting | Postoperative day 1
  The incidence of nausea and vomiting after surgery will be recorded
Baseline demographics | preoperatively
  Age, sex, body mass index (BMI), and comorbidities will be recorded
Blood Pressure | Blood pressure will be monitored continuously every 5 minutes and will be recorded prior to induction, post-induction, after the loading dose of dexmedetomidine, 4 hours and 12 hours postoperatively.
  Blood pressure (mmHg) will be monitored continuously every 5 minutes and will be recorded prior to induction, post-induction, after the loading dose of dexmedetomidine, 4 hours and 12 hours postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Main University Hospital, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No